CLINICAL TRIAL: NCT01092377
Title: The Effects of Iron and Omega-3 Fatty Acid Supplementation, Alone and in Combination, on Cognition, Immune System and Gut Microbiota: a Randomized, Double-blind, 2x2 Intervention Trial in Iron Deficient South African Children
Brief Title: The Effects of Iron and Omega-3 Fatty Acid Supplementation on Cognition and Immune Function in Iron Deficient Children
Acronym: FeFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North-West University, South Africa (Other)
Collaborators: Swiss Federal Institute of Technology (Other); Medical Research Council, South Africa (Other); Unilever R&D (Industry)
Responsible Party: Prof. Dr. Marius Smuts, North-West University, South Africa
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FeFA study 2010
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2010-12

CONDITIONS: Iron Deficiency; Anemia
MeSH Terms: conditions — Iron Deficiencies; Anemia | interventions — Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- DHA/EPA capsules and iron tablet (Experimental)
  Interventions: Dietary Supplement: DHA and EPA Fish Oil capsule; Dietary Supplement: Iron tablet
- DHA/EPA and placebo tablet (Experimental)
  Interventions: Dietary Supplement: DHA and EPA Fish Oil capsule; Other: Placebo tablet
- placebo capsules & placebo tablet (Placebo Comparator)
  Interventions: Dietary Supplement: Iron tablet; Other: Placebo tablet; Other: Placebo capsule
- iron tablet and placebo capsules (Experimental)
  Interventions: Other: Placebo capsule

INTERVENTIONS:
Dietary Supplement: DHA and EPA Fish Oil capsule — 2 DHA/EPA capsules on 4 days per week containing totally 420 mg DHA and 80 mg EPA, providing an average dose of 285.7 mg n-3 fatty acids per day
  Other Names: Provided by Burgerstein AG (Rapperswil, Switzerland)
  Arms: DHA/EPA and placebo tablet; DHA/EPA capsules and iron tablet
Dietary Supplement: Iron tablet — 1 iron tablet containing 50 mg of iron as ferrous sulfate will be administered on 4 days per week, providing an average iron dose of 28.6 mg iron per day.
  Other Names: Provided by Lomapharm (Paul Lohmann GmbH, Emmertal, Germany)
  Arms: DHA/EPA capsules and iron tablet; placebo capsules & placebo tablet
Other: Placebo tablet — Placebo tablet will be administered on 4 days per week and will be identical in appearance to the iron tablet.
  Other Names: Provided by Lomapharm (Paul Lohmann GmbH, Emmertal, Germany)
  Arms: DHA/EPA and placebo tablet; placebo capsules & placebo tablet
Other: Placebo capsule — Placebo capsules contain medium chain triglycerides and will be identical in appearance and total fat content to the DHA/EPA capsules.
  Other Names: Will be provided by R.P. Scherer GmbH (Eberbach, Germany)
  Arms: iron tablet and placebo capsules; placebo capsules & placebo tablet

SUMMARY:
The aim of this study is to determine if providing iron and a mixture of DHA and EPA, alone and in combination, to children with iron deficiency and poor n-3 fatty acid intake will improve their cognitive performance, activity levels and immune system.

Additionally, the effects on iron and fatty acid status, and gut microbiota, will be assessed.

DETAILED DESCRIPTION:
In populations of low socio economic status, such as found in South Africa, iron deficiency coexisting with a low intake of n-3 fatty acids could synergistically compromise both the intellectual performance and immune system of children.

Therefore, specific cognitive processes (domains) and specific immunization status markers and immune function modulators, that have been found to be affected by iron and n-3 fatty acid deficiency in children in previous studies will be assessed.

This will be the first human study that assesses the interactions of iron and n-3 fatty acid supplementation to iron deficient children in a two-by-two factorial, randomized, double-blind, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6-10 years
* Iron deficiency (Serum ferritin < 20 µg/L or zinc protoporphyrin > 70 µmol/mol heme in washed erythrocytes or TfR > 8.3 mg/L) with no or mild anaemia

Exclusion Criteria:

* Chronic illness
* Severe anemia (Hb < 80 g/L)
* Use of iron or n-3 fatty acid containing supplements

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in cognitive and behavioral performance and immune function | 8 months

SECONDARY OUTCOMES:
Change in activity levels, gut microbiota, iron status, fatty acid status and gene expression | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Marius Smuts, PhD, Study Director — North-West University; Michael B Zimmermann, PhD, Study Director — ETH Zürich; Linda Malan, MSc, Principal Investigator — North-West University; Jeannine Baumgartner, MSc, Principal Investigator — ETH Zürich
Locations (1):
- Valley of a Thousand Hills, Botha’s Hill, KwaZulu-Natal, South Africa

REFERENCES:
- [Derived] Malan L, Baumgartner J, Calder PC, Smuts CM. Low immune cell ARA and high plasma 12-HETE and 17-HDHA in iron-deficient South African school children with allergy. Prostaglandins Leukot Essent Fatty Acids. 2016 Jul;110:35-41. doi: 10.1016/j.plefa.2016.05.006. Epub 2016 May 13. PMID 27255641
- [Derived] Malan L, Baumgartner J, Zandberg L, Calder PC, Smuts CM. Iron and a mixture of DHA and EPA supplementation, alone and in combination, affect bioactive lipid signalling and morbidity of iron deficient South African school children in a two-by-two randomised controlled trial. Prostaglandins Leukot Essent Fatty Acids. 2016 Feb;105:15-25. doi: 10.1016/j.plefa.2015.12.005. Epub 2015 Dec 22. PMID 26869087
- [Derived] Malan L, Baumgartner J, Calder PC, Zimmermann MB, Smuts CM. n-3 Long-chain PUFAs reduce respiratory morbidity caused by iron supplementation in iron-deficient South African schoolchildren: a randomized, double-blind, placebo-controlled intervention. Am J Clin Nutr. 2015 Mar;101(3):668-79. doi: 10.3945/ajcn.113.081208. Epub 2014 Dec 31. PMID 25733652
- [Derived] Baumgartner J, Smuts CM, Malan L, Kvalsvig J, van Stuijvenberg ME, Hurrell RF, Zimmermann MB. Effects of iron and n-3 fatty acid supplementation, alone and in combination, on cognition in school children: a randomized, double-blind, placebo-controlled intervention in South Africa. Am J Clin Nutr. 2012 Dec;96(6):1327-38. doi: 10.3945/ajcn.112.041004. Epub 2012 Oct 24. PMID 23097272
- [Derived] Baumgartner J, Smuts CM, Aeberli I, Malan L, Tjalsma H, Zimmermann MB. Overweight impairs efficacy of iron supplementation in iron-deficient South African children: a randomized controlled intervention. Int J Obes (Lond). 2013 Jan;37(1):24-30. doi: 10.1038/ijo.2012.145. Epub 2012 Sep 4. PMID 22945607